CLINICAL TRIAL: NCT05506150
Title: Patient Important Gastrointestinal Bleeding in the ICU
Acronym: PIB
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: PIB_22
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Gastro Intestinal Bleeding; Patient Engagement; Family Members
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Patient Participation | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Interviews — Focused conversations to understand features of a GI bleed that are important to patients and families.
  Patients and family members are invited to participate in focused conversations. For interviews and focus groups, criterion sampling will be used. Investigators employed qualitative and quantitative methods to collect and analyze data. Quantitative data includes self-reported demographic characteristics of the patient and family members. Qualitative data about participants will be obtained through individual interviews and focused groups and project team field notes.

SUMMARY:
This study will engage patients and families to create a definition of what matters most to them about upper gastrointestinal (GI) bleeding. This information will help to define the outcome of "patient-important GI bleeding" which is a secondary endpoint for the ongoing international randomized trial REVISE (NCT03374800), comparing acid suppression versus no acid suppression in the intensive care unit (ICU). Other outcomes in REVISE are clinically important upper GI bleeding, mortality, pneumonia and Clostridioides difficile infection. Guided by patient and family input, a series of open-ended questions will elicit patient and family views about what matters most about this complication in interviews and focus groups. The investigators will develop the definition of "patient-important GI bleeding" by analyzing interview and focus group transcripts of critically ill survivors and family members of critically ill patients who may or may not have had GI bleeding, and who were not enrolled in the REVISE trial. Patient and family perspectives (anticipated to be different from what clinicians consider to be clinically important GI bleeding), will be used to refine a new trial outcome for research on GI bleeding in the intensive care unit (ICU). Also, study results will help clinicians understand how to better support patients and families; to explain testing and treatment options when GI bleeding occurs in practice in the ICU.

DETAILED DESCRIPTION:
This is a parallel mixed-methods multi-center study.

Design: This is a parallel mixed-methods multi-center study in which the qualitative data are dominant and patient and family involvement is paramount. Data collection will be quantitative and qualitative interviews and focus groups. The objective is to elicit views from patients and families regarding the features of a GI bleed that are important to patients. The investigators will recruit 6-10 patients and 6-10 family members for individual interviews, along with 6-10 focus groups consisting of 3-4 patients and family members.

ELIGIBILITY:
Patient Inclusion Criteria:

* Was admitted to an ICU, whether or not a GI bleed developed in the ICU
* > 18 years of age

Family Member Inclusion Criteria:

* Family members of ICU patients whose loved one was in the ICU for at least 72 hours, whether or not their family member developed a GI bleed
* > 18 years of age

Patient/Family Member Exclusion Criteria:

* Prohibitive communication challenges (e.g., serious psychological or psychiatric illness in the patient and/or family, inability of patient and/or family to communicate reasonably well in English or other languages for which an interpreter exists - professional staff or otherwise);
* Patient or family declines.
* Family member whose loved one died in ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been survived a stay in the ICU, and family members of critically ill patients.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of enrolment | Through study completion; an average of 1 year
  Enrolment will be deemed feasible when the following criteria are met: a) at least 15 surviving critically ill patients and 15 family members have been recruited; b) at least 8 focus groups have been completed; c) Representation of patients and families from several regions served by academic health sciences centres; 4) 80% participation rate for invited patients and families
GI Bleeding characteristics important to patients and families | Through study completion; an average of 1 year
  While clinically important GI bleeding is defined in research as bleeding accompanied by hemodynamic consequences, red blood cell transfusions or other invasive interventions, the concept of patient-important upper GI bleeding has not been developed for the ICU. In this study, the investigators will elicit views using open-ended questions about the tests and treatments about GI bleeding of greatest concern. This information will be analyzed inductively to develop and/or refine a new patient-centred definition of important bleeding. The investigators hypothesize that the GI bleed characteristics which are relevant to patients and families will not be the same as those relevant to clinicians. The inductive analysis involves the generation of categories and domains directly from the data, without pre-conceived notions of what these categories or domains might be.

CONTACTS AND LOCATIONS:
Locations (1):
- St Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Per the research ethics board-approved protocol, participants did not agree to data sharing (qualitative or quantitative)

REFERENCES:
- [Derived] Cook DJ, Swinton M, Krewulak KD, Fiest K, Dionne J, Debigare S, Guyatt G, Taneja S, Alhazzani W, Burns KEA, Marshall JC, Muscedere J, Gouskos A, Finfer S, Deane AM, Myburgh J, Rochwerg B, Ball I, Mele T, Niven D, English S, Verhovsek M, Vanstone M. What counts as patient-important upper gastrointestinal bleeding in the ICU? A mixed-methods study protocol of patient and family perspectives. BMJ Open. 2023 May 19;13(5):e070966. doi: 10.1136/bmjopen-2022-070966. PMID 37208143